CLINICAL TRIAL: NCT01042535
Title: A Phase 1/2 Study of Ad.p53 DC Vaccine in Combination With 1-methyl-D-tryptophan in Metastatic Solid Tumors and Invasive Breast Cancer
Brief Title: Vaccine Therapy and 1-MT in Treating Patients With Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-8461; NCI-2013-00516 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MCC-16025 (Other: H. Lee Moffitt Cancer Center and Research Institute); P30CA076292 (NIH)
Record Dates: First submitted 2010-01-04; First posted 2010-01-05 (Estimated); Results first posted 2015-03-05 (Estimated); Last update posted 2018-04-11 (Actual); Status verified 2018-03

CONDITIONS: Male Breast Cancer; Recurrent Breast Cancer; Stage IV Breast Cancer; Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: conditions — Breast Neoplasms, Male; Breast Neoplasms | interventions — Vaccines; 1-methyltryptophan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (vaccine therapy, 1-methyl-d-tryptophan) (Experimental): Participants receive adenovirus-p53 transduced dendritic cell (Ad.p53-DC) vaccine ID in weeks 1, 3, 5, and 10, and then every 3 weeks for 6 total doses. Participants also receive 1-methyl-d-tryptophan (indoximod) orally (PO) daily (QD) on days 1-21. Treatment with 1-methyl-d-tryptophan repeats every 28 days (patients with stable disease) for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: adenovirus-p53 transduced dendritic cell (DC) vaccine; Drug: 1-methyl-d-tryptophan; Other: Laboratory biomarker analysis

INTERVENTIONS:
Biological: adenovirus-p53 transduced dendritic cell (DC) vaccine — Given intradermally (ID)
  Other Names: Ad.p53-DC vaccine
Drug: 1-methyl-d-tryptophan — Given orally (PO)
  Other Names: indoximod; 1-MT
Other: Laboratory biomarker analysis — Correlative studies

SUMMARY:
This randomized phase I/II trial studies the side effects and best dose of vaccine therapy and to see how well it works when given together with 1-methyl-D-tryptophan (1-MT) in treating patients with metastatic breast cancer. Vaccines made from a person's tumor cells and white blood cells may help the body build an effective immune response to kill tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) and safety using Common Terminology Criteria for Adverse Events (CTCAE) version 4.0, of the combination Ad.p53 DC vaccine (adenovirus-p53 transduced dendritic cell vaccine) plus 1-MT in patients with any solid malignancy that has mutated p53 by immunohistochemistry (IHC). (Phase I) II. To determine efficacy (objective response rate) of the combination Ad.p53 DC vaccine plus 1-MT in metastatic breast cancer patients whose tumor expresses mutated p53 by IHC. (Phase II)

SECONDARY OBJECTIVES:

I. To collect preliminary data on and study the p53 specific interferon-gamma (IFN-gamma) enzyme-linked immunosorbent spot (ELISPOT) measurement at baseline, week 7 and week 16. (Phase I) II. To collect preliminary data on and study the percentage of p53 specific IFN-gamma ELISPOT responders at week 7 and 16. (Phase II) III. To collect preliminary data on and study progression-free survival on the study treatment. (Phase II) IV. To collect preliminary data on and study response and progression-free survival on the subsequent chemotherapy if administered. (Phase II) V. To collect preliminary data on and study the effects of 1-methyl-D-tryptophan (1-MT) on serum kynurenine, serum tryptophan, C reactive protein, and circulating T-regulatory cells (clusters of differentiation (CD)4+ 25+ CD127low forkhead box P3+ (FoxP3+)) by flow cytometry at each vaccination point on study when compared their corresponding baseline. (Phase II)

OUTLINE: This is a phase I, dose escalation study followed by a phase II study.

Patients receive adenovirus-p53 transduced dendritic cell vaccine intradermally (ID) in weeks 1, 3, 5, and 10, and then every 3 weeks for 6 total doses. Patients also receive 1-methyl-d-tryptophan orally (PO) once daily (QD) on days 1-21. Treatment with 1-methyl-d-tryptophan repeats every 28 days (patients with stable disease) for up to 12 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* In the phase I patients with any solid tumor positive for p53 by IHC (>= 5% of cells with any degree of nuclear staining) staining; for the phase II, patients must have histologically or cytologically confirmed metastatic invasive breast cancer that is positive for p53 staining by IHC (>= 5% of cells with any degree of nuclear staining); patients will sign a separate consent for the p53 testing, and those that meet the above requirements will then be allowed to sign the vaccine trial consent
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 20 mm with conventional techniques or as >= 10 mm with spiral computed tomography (CT) scan
* There are no restrictions on prior therapies for the phase I part of the trial; for the phase II, patients may have received up to 2 prior lines of chemotherapy (not counting endocrine therapy lines) with the last dose of chemotherapy given 3 weeks (6 weeks for nitrosoureas and mitomycin C) prior to initiation on this study
* Life expectancy of greater than 4 months
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (Karnofsky >= 70%)
* Leukocytes >= 3,000/μL
* Absolute neutrophil count >= 1,500/μL
* Platelets >= 100,000/μL
* Total bilirubin within normal institutional limits unless patient has Gilbert's disease
* Aspartate aminotransferase (AST) /serum glutamic oxaloacetic transaminase (SGOT) /alanine aminotransferase (ALT) /serum glutamic pyruvate transaminase (SGPT) =< 2.5 X institutional upper limit of normal
* Creatinine within normal institutional limits OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Thyroid-stimulating hormone (TSH), luteinizing hormone (LH), follicle-stimulating hormone (FSH), adrenocorticotropic hormone (ACTH) showing normal pituitary function; these values may deviate if in the opinion of the investigator these are normal pituitary responses to another endocrine condition such as suboptimally treated hypothyroidism
* Patients with known brain metastases will only be eligible after their tumors have been treated with definitive resection and/or radiotherapy and they are neurologically stable for at least 1 month off steroids
* No history of gastrointestinal disease causing malabsorption or obstruction such as but not limited to Crohn's disease, celiac sprue, tropical sprue, bacterial overgrowth/blind loop syndrome, gastric bypass surgery, strictures, adhesions, achalasia, bowel obstruction, or extensive small bowel resection
* Sexually active women of child-bearing potential must agree to use two forms of contraception (hormonal and barrier method of birth control or abstinence) prior to study entry and for the duration of study participation; males should use barrier contraception or abstinence during the study; use of contraception or abstinence should continue for a minimum of 1 month after completion of the study; should a woman become pregnant or suspect she is pregnant while participating in this study, she should discontinue the study drug and inform her treating physician immediately; a pregnancy test is required prior to study enrollment and monthly while on treatment with 1-MT for all women of child-bearing potential; also men should be discouraged from fathering children while on treatment
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 3 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 3 weeks earlier
* Patients may not receive any other investigational agents or chemotherapy to treat their underlying malignancy while on study; patients who are stable on prior endocrine therapies (i.e. aromatase inhibitors, tamoxifen, and fulvestrant) may stay on these treatments
* Patients with known untreated brain metastases are excluded from this clinical trial; patients with stable previously treated lesions in a patient off steroids and radiation for 1 month are not excluded
* History of allergic reactions (significant urticaria, angioedema, anaphylaxis) attributed to compounds of similar chemical or biologic composition to 1-methyl-D-tryptophan; this would include L-tryptophan or 5-hydroxy-tryptophan supplements
* No supplements containing L-tryptophan or derivatives thereof are allowed to be taken while on study; also ingestion of antacid compounds should be timed a minimum of 2 hours before or after ingestion of 1-MT
* Patients with any active autoimmune disease (i.e. psoriasis, extensive atopic dermatitis, asthma, inflammatory bowel disease ([IBD), multiple sclerosis (M.S.), uveitis, vasculitis), chronic inflammatory condition, or any condition requiring concurrent use of any systemic immunosuppressants or steroids for any reason would be excluded from the study; any patient with an allo-transplant of any kind would be excluded as well; this would include those with a xenograft heart valve to avoid the potential risk of any immune reaction causing valvular degeneration; mild-intermittent asthma requiring only occasional beta-agonist inhaler use or mild localized eczema will not be excluded
* Uncontrolled concurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, myocardial infarction or percutaneous coronary interventions within the last 6 months, cardiac arrhythmia, active autoimmune diseases, or major psychiatric illness/social situations that would limit compliance with study requirements as judged by the primary investigator at each site; those with well controlled, chronic medical conditions under the supervision of the patient's primary physician (i.e. hypertension, hyperlipidemia, coronary heart disease, diabetes mellitus) would not be excluded
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with 1-methyl-D-tryptophan
* Human immunodeficiency virus (HIV)-positive patients and those with other acquired/inherited immunodeficiencies are ineligible
* Patients with more than one active malignancy at the time of enrollment
* Patients who have received any prior experimental active immunotherapy consisting of targeted monoclonal antibodies or pharmaceutical compounds are excluded; prior experimental vaccine patients may be enrolled if approved by the principal investigator (PI); patients who have received commercially available active immunotherapies such as adjuvant interferon must have completed therapy over 1 year prior to enrollment and have no evidence of autoimmune sequelae; prior therapy with approved monoclonal antibodies such as bevacizumab, cetuximab, panitumumab, or trastuzumab is allowed; concurrent treatment with these agents and the study treatment is not allowed
* Human epidermal growth factor receptor 2 positive (HER2+) patients (IHC 3+ and/or fluorescent in situ hybridization [FISH] HER2/centromere portion of chromosome 17 [CEP17] ratio > 2) who require treatment with trastuzumab or lapatinib are not eligible for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2009-12-28 (Actual); Primary Completion 2014-12-01 (Actual); Study Completion 2018-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hatem Soliman, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at Moffitt Cancer Center from December 28, 2009, through February 11, 2014.
Period: Overall Study
Arm/Group | Treatment (Vaccine Therapy, 1-methyl-d-tryptophan)
Started | 44
Completed | 36
Not Completed | 8
Not completed — disease progression prior to treatment | 3
Not completed — disease progression during treatment | 3
Not completed — complications from other disease | 2

BASELINE CHARACTERISTICS:
Population: All participants
Arm/Group | Treatment (Vaccine Therapy, 1-methyl-d-tryptophan)
Number analyzed (Participants) | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 36
  >=65 years | 8
Age, Continuous [Mean (Full Range); unit: years] | 52.68 [27 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 44

OUTCOME MEASURES:

1. Primary Outcome: Phase 1 - Maximum Tolerated Dose (MTD) in Milligrams (mg)
Description: MTD of 1-methyl-d-tryptophan (indoximod) given by mouth (PO), twice a day (BID), with up to 6 fixed doses Ad.p53 DC vaccinations every 2 weeks (q2wks). This phase 1 study used a 3+3 design with 7 indoximod dose levels (DL) (100 mg, 200 mg, 400 mg, 800 mg daily (QD) then 800 mg, 1,200 mg, and 1,600 mg PO BID +up to 6 fixed dose Ad.p53 DC vaccinations q2wks. Toxicity was assessed according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v4.0. The MTD is the highest dose level below the maximally administered dose (MAD) that is safely tolerated among 6 treated patients, that is, 0 or 1 out of 6 patients experiences a dose limiting toxicity (DLT).
Time Frame: Up to 4 weeks
Population: Phase I Participants who Received at Least 1 Dose of Ad.p53DC+indoximod
Measure: Number; unit: indoximod dose in mg
Arm/Group | Treatment (Vaccine Therapy, 1-methyl-d-tryptophan)
Number analyzed (Participants) | 30
indoximod dose in mg | 1600

2. Primary Outcome: Phase 2 - Number of Participants With Stable Disease In Response to Study Therapy
Description: Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.
Time Frame: Up to 16 weeks
Population: All evaluable participants at time of analysis
Measure: Number; unit: participants
Arm/Group | Treatment (Vaccine Therapy, 1-methyl-d-tryptophan)
Number analyzed (Participants) | 21
participants | 4

3. Secondary Outcome: Phase 1 - Number of Participants With Objective Response at 6 Weeks
Description: Immunologic Response defined as Interferon-γ (IFN-γ) p53 T cell specific enzyme-linked immunospot (ELISPOT) assay count Summarized using both point estimates and the 95% exact confidence intervals based on the binomial distribution. Briefly, 2x10^5 mononuclear cells obtained from the peripheral blood of patients will be plated in quadruplicates in 96-well multiscreen mixed cellulose ester (HA) filtration plates, processed and incubated, spots will be visualized. The number of spots will be calculated per 10^6 cells. Untreated peripheral blood mononuclear cells (PBMNC) will represent a negative control and PBMNC stimulated with 10 µg/ml Concanavalin A (ConA) - positive control.
Time Frame: At 6 weeks
Population: Phase I Participants who Received at Least 1 Dose of Ad.p53DC+indoximod
Measure: Number; unit: participants
Arm/Group | Treatment (Vaccine Therapy, 1-methyl-d-tryptophan)
Number analyzed (Participants) | 30
participants | 0

4. Secondary Outcome: Phase 2 - Number of Participants With Clinical Benefit From Chemotherapy After Vaccination
Description: Clinical response rate evaluated using the Response Evaluation Criteria in Solid Tumors (RECIST) criteria. Complete Response (CR): Disappearance of all target lesions. Partial Response (PR): At least a 30% decrease in the sum of the diameter (LD) of target lesions, taking as reference the baseline sum LD. Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.
Time Frame: Up to 3 years
Population: All evaluable participants at time of analysis
Measure: Number; unit: participants
Arm/Group | Treatment (Vaccine Therapy, 1-methyl-d-tryptophan)
Number analyzed (Participants) | 21
participants
  Complete Response (CR) | 1
  Partial Response (PR) | 7
  Stable Disease (SD) | 2

5. Secondary Outcome: Phase 2 - Median Progression Free Survival (PFS) in Weeks
Description: Progressive Disease (PD): Appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions. PFS: Time from study entry to documentation of radiologic progressive disease or death, assessed up to 3 years.
Time Frame: Up to 3 years
Population: All evaluable participants at time of analysis
Measure: Median (Full Range); unit: weeks
Arm/Group | Treatment (Vaccine Therapy, 1-methyl-d-tryptophan)
Number analyzed (Participants) | 21
weeks | 6.85 [3.8 to 18.1]

6. Other Pre Specified Outcome: Phase 2 - Change in Biomarker Level
Description: Biomarkers include serum kynurenine, serum tryptophan, C reactive protein, and circulating T-regulatory cell levels (CD4+ 25+ CD127low forkhead box protein 3+ (FoxP3+). Appropriate t-tests and/or Wilcoxon test will be employed to study changes over time.
Time Frame: Baseline to week 16
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 4 years, 3 months
Description: Only 41 of 44 enrolled were at risk. 3 participants had disease progression prior to treatment.
Arm/Group | Treatment (Vaccine Therapy, 1-methyl-d-tryptophan)
Serious Adverse Events (participants affected / at risk) | 14/41
Other Adverse Events (participants affected / at risk) | 37/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Vaccine Therapy, 1-methyl-d-tryptophan) (N=41)
Anemia (Blood and lymphatic system disorders) | 1 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Eye disorders - Other, Visual disturbance (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Skin infection (Infections and infestations) | 2 (2)
Alkaline phosphatase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Neoplasms benign - Other, Disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Nervous system disorder - Other, Disease progression (Nervous system disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Vaccine Therapy, 1-methyl-d-tryptophan) (N=41)
Fatigue (General disorders) | 27 (39)
Edema limbs (General disorders) | 5 (5)
Fever (General disorders) | 3 (4)
Flu like symptoms (General disorders) | 2 (2)
Pain (General disorders) | 2 (3)
Anorexia (Metabolism and nutrition disorders) | 14 (16)
Hyperglycemia (Metabolism and nutrition disorders) | 13 (20)
Hypoalbuminemia (Metabolism and nutrition disorders) | 10 (14)
Hyponatremia (Metabolism and nutrition disorders) | 7 (9)
Dehydration (Metabolism and nutrition disorders) | 4 (4)
Hyperkalemia (Metabolism and nutrition disorders) | 3 (4)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (4)
Hypokalemia (Metabolism and nutrition disorders) | 3 (4)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2)
Alkaline phosphatase increased (Investigations) | 14 (20)
Aspartate aminotransferase increased (Investigations) | 12 (19)
Lymphocyte count decreased (Investigations) | 11 (16)
Alanine aminotransferase increased (Investigations) | 8 (11)
White blood cell decreased (Investigations) | 8 (10)
Neutrophil count decreased (Investigations) | 5 (5)
Platelet count decreased (Investigations) | 3 (5)
Creatinine increased (Investigations) | 2 (2)
Nausea (Gastrointestinal disorders) | 15 (17)
Constipation (Gastrointestinal disorders) | 9 (10)
Vomiting (Gastrointestinal disorders) | 10 (13)
Abdominal pain (Gastrointestinal disorders) | 8 (8)
Diarrhea (Gastrointestinal disorders) | 7 (7)
Dry mouth (Gastrointestinal disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Toothache (Gastrointestinal disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (9)
Bone pain (Musculoskeletal and connective tissue disorders) | 6 (8)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 4 (5)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Anemia (Blood and lymphatic system disorders) | 15 (32)
Hemolysis (Blood and lymphatic system disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 10 (12)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Headache (Nervous system disorders) | 8 (8)
Peripheral sensory neuropathy (Nervous system disorders) | 7 (9)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2)
Urinary tract infection (Infections and infestations) | 3 (3)
Hypotension (Vascular disorders) | 2 (2)
Breast pain (Reproductive system and breast disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes